CLINICAL TRIAL: NCT00240279
Title: The Effect of Rosuvastatin on Aortic Stiffness in Hemodialysis Patients in the AURORA Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4522IL/0096 Dutch SubStudy; D3562C00096
Record Dates: First submitted 2005-10-16; First posted 2005-10-18 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Hypercholesterolemia
Keywords: high blood cholesterol levels
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin
Procedure: aortic pulse wave velocity measurements

SUMMARY:
To investigate the effect of rosuvastatin compared to placebo on the aortic stiffness in hemodialysis patients as measured by pulse wave velocity (at 3, 6 and 12 months)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, between 50 and 80 years of age, end stage renal failure patients receiving hemodialysis

Exclusion Criteria:

* Received statins within past 6 months, a clear indication for use of lipid altering drug, contra indication for lipid altering drug, history of statin induced myopathy items in very

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of rosuvastatin compared to placebo on the aortic stiffness in hemodialysis patients as measured by pulse wave velocity (at 3, 6 and 12 months)

SECONDARY OUTCOMES:
To investigate the effect of rosuvastatin compared to placebo on the aortic pressure wave in hemodialysis patients (at 3 months/ 6 months and 12 months).

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Crestor Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Nieuwegein, Netherlands